CLINICAL TRIAL: NCT05262933
Title: Effect of Preoperative Coffee Consumption on Intraoperative and Post Operative Outcomes in Cesarean Section With Spinal Anesthesia
Brief Title: Effects of Preoperative Coffee Consumption in Cesarean Sections Under Spinal Anesthesia
Status: Completed | Type: Observational
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Gamze Talih, Associate Professor, TC Erciyes University
Other Study IDs: 2021/825
Record Dates: First submitted 2022-02-21; First posted 2022-03-02 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Hypotension After Spinal Anesthesia; Post-Dural Puncture Headache
MeSH Terms: conditions — Post-Dural Puncture Headache | interventions — Coffee; Water

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- coffee (n= 70): Patients are planned to drink brewed coffee 2 hours before surgery.
  Interventions: Other: coffee
- control (n=70): Patients are planned to drink water 2 hours before surgery.
  Interventions: Other: Water

INTERVENTIONS:
Other: coffee — It will be given to patients brewed coffee to drink and evaluated to hypotension and post spinal puncture headache
  Other Names: It will be given to patients brewed coffee to drink
  Groups: coffee (n= 70)
Other: Water — It will be given to patients water to drink and evaluated to hypotension and post spinal puncture headache
  Other Names: It will be given to patients water to drink
  Groups: control (n=70)

SUMMARY:
The prospective study is planned in a university hospital. Spinal anesthesia is widely used for cesarean section currently for its safety, low cost, reliability, easiness to administer, immediate effect, and well-operating conditions. However spinal anesthesia has some complications as hypotension, bradycardia and Post Dural Puncture Headache (PDPH). A practical strategy for avoiding hypotension during initiation of spinal anesthesia for cesarean delivery includes intravenous crystalloid, in conjunction with administration of vasopressors. PDPH is one of the most frequent complications of spinal anesthesia. Conservative therapies such as bed rest, hydration, and caffeine are commonly used as management. For this study, coffee group of patients will be given unsweetened brewed coffee 150 ml until 2-4 hours before surgery. Patients who accept to drink brewed coffee ( coffee group) and water( control group) will be included in the study. The patient's heart rate, blood pressure, oxygen saturation will be monitored and recorded during operation. Intraoperative will be recorded to amount of vasopressor and intraveous crystalloid. Whether the patient develops PDPH in the postoperative period will be followed for 3 days. In addition abdominal auscultation for bowel sounds hourly and the time of first bowel movements will be recorded. According to the patient's statement, the time of first flatulence and defecation will be followed and recorded.

ELIGIBILITY:
Inclusion Criteria:

* patients who accept to participate in the study
* patient who limit the consumption of caffeinated beverages such as coffee and tea during pregnancy
* Patients with known caffeine or coffee allergy

Exclusion Criteria:

* patients who refuse to participate in the study
* Patients with known cardiovascular disease
* Patients with known cerebrovascular disease
* patients with known neurological, neurodegenerative or psychiatric disease
* patients with known liver failure
* patient followed up with eclampsia and preaclampsi
* higher number of needle passes in spinal anesthesia
* patients treated with an antiemetic

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: parturient women aged 18-45
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
hypotension | intraoperative time period
  effects of orally coffee intake on spinal anesthesia induced hypotension

SECONDARY OUTCOMES:
Post-dural puncture headache | post operative 3 days
  Effects of orally coffee intake on postdural puncture headache
intestinal motility, first flatus | post operative 3 days
  Effects of orally coffee intake on postoperative intestinal motility

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University, Kayseri, Turkey (Türkiye)